CLINICAL TRIAL: NCT01486199
Title: Imaging Airway Liquid Absorption in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Tim Corcoran, Assistant Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1R01HL108929-01 (NIH); R01HL108929 (NIH)
Record Dates: First submitted 2011-11-18; First posted 2011-12-06 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; mucociliary clearance; airway surface liquid; nuclear medicine
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CF pediatric (Experimental): In the pediatric arm 10 CF subjects ages 6-14 will perform absorptive clearance scans at baseline and at t=2 years.
  Interventions: Other: Absorptive clearance scan
- Controls adult (Experimental): In the adult control arm 10 healthy adult subjects will perform a single absorptive clearance scan.
  Interventions: Other: Absorptive clearance scan

INTERVENTIONS:
Other: Absorptive clearance scan — Subjects will inhale a nebulized mixture of the radiopharmaceuticals Indium 111-DTPA and Technetium 99m-sulfur colloid.

SUMMARY:
The investigators are developing a new nuclear medicine imaging technique for measuring liquid absorption in the airways that can be applied to screen new medications being developed to treat cystic fibrosis (CF). The investigators believe that the absorption of the small molecule radiopharmaceutical Indium 111-diethylenetriaminepentaacetic acid (In-DTPA) will indicate changes in liquid absorption in the airways and demonstrate whether new CF medications will be effective. In this study the investigators will further develop this technique through testing involving pediatric CF patients and healthy control subjects.

DETAILED DESCRIPTION:
The investigators have recently developed a novel aerosol-based imaging technique to detect changes in liquid absorption in the airways - a central pathophysiological process known to be important in cystic fibrosis (CF) lung disease. This technique may provide a measure of disease severity and indication of therapeutic correction in advance of currently available outcome measures. It involves the simultaneous delivery of two radiopharmaceuticals by inhalation: one an absorbable small-molecule (Indium-111 labeled diethylenetriaminepentaacetic acid; In-DTPA) and the other a non-absorbable particle (Technetium 99m labeled sulfur colloid; Tc-SC). The overarching hypothesis is that In-DTPA absorption provides a quantifiable, non-invasive measurement of airway liquid absorption that (a) is sensitive to CF genotype, (b) uniquely identifies basic disease phenotype and predicts disease severity, and (c) is modulated by therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy control arm:

  * subjects 18 years old or older without a diagnosis of lung disease.
* Pediatric CF arm:

  * subjects 6-14 years with a diagnosis of cystic fibrosis as determined by sweat test or genotype
  * subjects who are clinically stable as determined by the pediatrician co-investigator
  * subjects must have a previously demonstrated ability to perform reproducible pulmonary function testing based on previous clinical visits.
* Females in all groups who are of child-bearing potential will need to have a negative urine pregnancy test.

Exclusion Criteria:

* Adult healthy control arm:

  * FEV1%p < 80% of predicted
  * nursing mother
  * positive urine pregnancy test or unwilling to test
  * cigarette smoker (regular smoking within 6 months of study).
* Pediatric CF arm:

  * FEV1%p < 40% of predicted
  * nursing mother
  * positive urine pregnancy test for females of childbearing potential
  * unable or unwilling to comply with test procedure
  * cigarette smoker (regular smoking within 6 months of study).
  * Subjects unable to lie recumbent without moving for the 80 minute imaging period will be excluded.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Corcoran, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Locke LW, Myerburg MM, Weiner DJ, Markovetz MR, Parker RS, Muthukrishnan A, Weber L, Czachowski MR, Lacy RT, Pilewski JM, Corcoran TE. Pseudomonas infection and mucociliary and absorptive clearance in the cystic fibrosis lung. Eur Respir J. 2016 May;47(5):1392-401. doi: 10.1183/13993003.01880-2015. Epub 2016 Mar 23. PMID 27009167
- [Derived] Locke LW, Myerburg MM, Markovetz MR, Parker RS, Weber L, Czachowski MR, Harding TJ, Brown SL, Nero JA, Pilewski JM, Corcoran TE. Quantitative imaging of airway liquid absorption in cystic fibrosis. Eur Respir J. 2014 Sep;44(3):675-84. doi: 10.1183/09031936.00220513. Epub 2014 Apr 17. PMID 24743971

RESULTS

PARTICIPANT FLOW:
Groups:
- CF Pediatric: Cystic Fibrosis subjects ages 6-14
- Controls Adult: Adult control subjects 18 or older
Period: Baseline Study Day
Arm/Group | CF Pediatric | Controls Adult
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Period: Two Year Period Between Study Days
Arm/Group | CF Pediatric | Controls Adult
Started | 10 | 0
Completed | 9 | 0
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Study Day at t= 2 Years
Arm/Group | CF Pediatric | Controls Adult
Started | 9 | 0
Completed | 9 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CF Pediatric | Controls Adult | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.5 (1.5) | 31.2 (15.0) | 20.9 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Absorptive Clearance Rate
Description: Absorptive clearance rate measured 80 minutes after radiopharmaceutical inhalation. Absorptive clearance is the absorptive component of the clearance of Indium 111-diethylenetriaminepentaacetic acid (In-DTPA) from the lungs.
Time Frame: study day 1
Population: One pediatric subject did not deposit sufficient aerosol to be analyzed. One control subject did not perform imaging procedures after signing consent because of a low result on a screening pulmonary function testing.
Measure: Mean (Standard Deviation); unit: percent cleared / 80 minutes
Groups:
- CF Pediatric: CF subjects ages 6-14
Arm/Group | CF Pediatric | Controls Adult
Number analyzed (Participants) | 9 | 9
percent cleared / 80 minutes | 34.0 (10.4) | 17.7 (6.9)
Statistical Analysis 1: Comparison: CF Pediatric vs Controls Adult; Comparing absorptive clearance in CF children vs adult controls; Test type: Equivalence — alpha=0.05; p = 0.002, t-test, 2 sided

2. Primary Outcome: Mucociliary Clearance Rate
Description: Mucociliary clearance rate measured 80 minutes after radiopharmaceutical inhalation. Mucociliary clearance rate is the rate of clearance of Technetium sulfur colloid (Tc-SC) from the lungs.
Time Frame: study day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent cleared / 80 minutes
Arm/Group | CF Pediatric | Controls Adult
Number analyzed (Participants) | 9 | 9
percent cleared / 80 minutes | 22.8 (13.7) | 31.4 (13.1)
Statistical Analysis 1: Comparison: CF Pediatric vs Controls Adult; Comparison of mucociliary clearance in CF children compared to healthy adults; Test type: Equivalence — alpha = 0.05; p = 0.20, t-test, 2 sided

3. Secondary Outcome: Absorptive Clearance Rate
Description: Absorptive Clearance Rate measured 80 minutes after radiopharmaceutical inhalation. Absorptive clearance is the absorptive component of the clearance of In-DTPA from the lungs.
Time Frame: t=2 years
Population: Only pediatric CF subjects performed 2 year follow-up scan. One subject did not perform the second imaging day since day one image quality was poor. Two other subjects had poor imaging data on follow up day and were therefore not included in analysis.
Measure: Mean (Standard Deviation); unit: percent cleared / 80 min
Arm/Group | CF Pediatric | Controls Adult
Number analyzed (Participants) | 7 | 0
percent cleared / 80 min | 28.6 (9.9) |
Statistical Analysis 1: Comparison: CF Pediatric; Comparing absorptive clearance at t=0 vs t=2 years in pediatric CF subjects; Test type: Equivalence — alpha=0.05; p = 0.24, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Mucociliary Clearance Rate
Description: as for outcome 2
Time Frame: t=2 years, measure made 80 minutes after radiopharmaceutical inhalation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent cleared / 80 minutes
Arm/Group | CF Pediatric | Controls Adult
Number analyzed (Participants) | 7 | 0
percent cleared / 80 minutes | 22.0 (13.1) |
Statistical Analysis 1: Comparison: CF Pediatric; Comparing mucociliary clearance at t=0 and t=2yrs in pediatric CF subjects; Test type: Equivalence — alpha=0.05; p = 0.87, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Groups:
- Controls Adult: adult controls 18 or older
Arm/Group | CF Pediatric | Controls Adult
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes